CLINICAL TRIAL: NCT04102969
Title: Effectiveness of Benson Relaxation Technique on Perceived Stress and Pain Among Hemodialysis Patients in an Urban Community Amman, Jordan: a Randomized Trial
Brief Title: Benson Relaxation Technique on Perceived Stress and Pain Among Hemodialysis Patients
Acronym: BRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Haya Ibrahim Abu Maloh, PhD Nursing Student, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JKEUPM-2019-340
Record Dates: First submitted 2019-09-16; First posted 2019-09-25 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Relaxation
Keywords: Benson relaxation; Benson response; Relaxation response

STUDY DESIGN:
Intervention Model Description: A cluster randomized controlled trial design (RCT) with two conditions (experimental versus control group) and four repeated measures time points for this study; at baseline test (before intervention), a post-test (immediately after the intervention), and follow up at one month post-intervention, and follow up at two months' post-intervention.
  Two hospitals will be divided in to Experimental and control hospital. participants in the experimental hospital will receive the intervention of Benson Relaxation technique (Intervention group).
  participants in the control hospital will receive the nutrition package session (control group).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinding will be used in this study, by not telling the participants, interventionist, and research assistants what the researcher is looking for to study, what the research outcomes are, and by making them not aware who is receiving the intervention or in which group they are in control or intervention group. So, the participants, interventionist, and research assistants who are in the study will be less likely to inadvertently bias the result.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group will be instructed by an interventionist who is qualified in stress management and relaxation will perform the Benson relaxation technique to the intervention group to perform the Benson relaxation technique two times a day for 10 minutes during the study period ( two months).
  Training session of the technique will be repeated if necessary over one or two sessions until the interventionist confirm that the participants acquired sufficient skills. A total of two hours will be scheduled for each session and will be coordinated with the nursing manager of the hemodialysis department.
  Interventions: Behavioral: Benson Relaxation Technique
- Control Group (Other): A qualified nutritionist will run out a nutrition package session for hemodialysis patients in the control group. This nutrition package session will be for one session for one hour.
  Interventions: Other: Nutrition Package Session

INTERVENTIONS:
Behavioral: Benson Relaxation Technique — Benson relaxation technique will be performed two times a day for 10 minutes during the study period ( two months) for the intervention group.
  Arms: Intervention group
Other: Nutrition Package Session — A nutrition package session will be given to the control group.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the effectiveness of Benson relaxation technique on perceived stress and pain among hemodialysis patients at governmental hospitals in Amman, Jordan. Half of the participants the intervention group will receive the intervention of Benson relaxation technique, while the other half the control group will receive a nutrition package session.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of Benson relaxation technique on perceived stress and pain among hemodialysis patients at governmental hospitals in Amman, Jordan at baseline, post-test, one and two months' follow-up assessment.

Two large governmental hospitals in Amman, Jordan will be randomly assigned in to experimental hospital (n=1) and control hospital (n=1). One hundred hemodialysis patients will be randomly assigned to experimental group (n = 50) and control group (n = 50). Intervention group will receive the Benson relaxation technique and the control group will receive a nutrition session. Measures of Perceived stress and pain using the Perceived stress scale (PSS) and the Short-Form McGill Pain Questionnaire (SF-MPQ) will be administered at pre-test, post-test, one and 2-months follow-up assessment. Data collection will be performed by two research assistance who are blind to treatment conditions.

Sample size:

The sample size for this study will be calculated to achieve a power of 0.80 with an alpha significance of 0.05 (2-tailed). The sample size for hemodialysis patients is based on a previous intervention study.

The following is sample size calculation formula:

n = (Z1-α/2+Z1-β)2 ×2×σ2 (µ1- µ2)2 σ² = (n1 -1) σ 12+ (n2-1) σ 22 (n1+n2)-2 Where, n1 = 44, σ1= 2.75, and the µ1= 11.52 before the intervention, and n2= 44, σ2 = 2.13 and the µ2 = 10.22 after the intervention (Davanloo & Heidarigorji, 2014).

σ² = (44 -1) 4.02+ (44-1) 4.222 (44+44)-2 σ² = 688+ 765.7612 86 σ² = 1453.7612 86 σ² = 16.9042 n= (1.96+0.84)2 ×2×16.9042 (16.10-13.11)2 n= 7.851204 ×2×16.0497 8.9401

n= 265.4366453 8.9401

n= 29.6902344 n= 30 for each group The study will use cluster randomized controlled trials design to achieve power of the study (DEFF) estimated to be 1.3.

n = 1.3 x 30= 39 n=39 With considering 20% attrition rate= 39/0.8= 48.75. The total sample size is n= 100. Each group will have 50 participants. Each cluster will have 50 participants.

Intervention group:

Intervention group will be instructed to perform the Benson relaxation technique two times a day for 10 minutes during the study period as follows:

Training sessions:

An interventionist who is qualified in stress management and relaxation will perform the Benson relaxation technique to the intervention group. The training sessions will be conducted before dialysis session in a warm quite room with efficient light, temperature, and ventilation in the hemodialysis department. The interventionist will first teach the participants how to perform deep breathing, the interventionist will teach the participants the 334 deep breathing technique for 5 minutes. Then the interventionist will verbally describe the Benson's relaxation technique for the eligible participants. Patient will also be instructed to perform the Bensons Relaxation Technique according to the following steps:

1. Sit quietly in a comfortable position.
2. Close your eyes.
3. Deeply relax all your muscles, beginning at your feet, progressing up to your face, and keep them deeply relaxed.
4. Breathe through your nose. Become aware of your breathing. As you breathe out, say the word 'one' silently to yourself. For example, breath in . . . out, 'one'; in . . . out, 'one'; etc.
5. Continue for 10 min. You may open your eyes to check the time, but do not use an alarm. When you ﬁnish, sit quietly for several minutes at ﬁrst with closed eyes and later with opened eyes.
6. Do not worry about whether you are successful in achieving a deep level of relaxation. Maintain a passive attitude and permit relaxation to occur at its own pace. When distracting thoughts occur, ignore them and continue repeating 'one'. With practice, the response should come with little effort. Practice the technique twice a day, but not within 2 h after any meal as the digestive processes seem to interfere with the elicitation of anticipated changes.

Then, the participants will watch a video of Benson relaxation technique and perform it in the presence of the interventionist who will provide a feedback by evaluating the participants' skills in performing the technique. After the training session, the participants will be asked to practice it twice a day for the next two days. Then, the participant will perform the technique in the presence of the interventionist in order to ensure that they have acquired sufficient skills. The technique will be repeated if necessary over one or two sessions until the interventionist confirm that the participants acquired sufficient skills. A total of two hours will be scheduled for each session and will be coordinated with the nursing manager of the hemodialysis department.

A Compact disc (CD) on the relaxation technique will be given to the patients enable to ensure their effective learning. They will be asked to listen to the Compact disc (CD) only twice a day at home and simultaneously perform the technique for 10 min for eight weeks. If performing the technique for the participants should be done twice a day at two specific times with 7-8-hour interval between each episode. The participants will be emphasized not to forget to perform the technique. However, if it happened, they will be asked to do it as soon as possible.

To ensure the participants compliance with Benson relaxation technique:

The video of Benson relaxation technique will be displayed in hemodialysis sessions during the study period to remind the participants to perform Benson relaxation technique. Whenever the participants have hemodialysis session, they will be performing the first time during the session and the second time will be at home.

Also, a self-reporting "performance record from" will be daily filled out by the participants to ensure their compliance with Benson's relaxation technique. Every week, the interventionist will be referring to the hemodialysis unit and will be encouraging the participants to perform the technique and at the same time, their "performance record forms" will be collected. Moreover, to ensure that the participants underwent the intervention appropriately, the participants will perform the technique again in the presence of the interventionist. Additionally, the interventionist will do a recall sheet and ask the family member who accompany the participants during hemodialysis sessions to ensure the participants compliance with Benson relaxation technique.

The interventionist will take the contact information and number of the participants and the family member that accompany the participant and keep it in a coding book separately. Then interventionist will make a group on Whats App for all the participants and send them the Benson relaxation technique video twice a day in specific times to remind the participants to perform the technique. Also, the interventionist will make a group on Whats App for the family member who accompany the participant during the hemodialysis session and send them a kind reminder as they can remind the participant to perform Benson relaxation technique.

Furthermore, the identification card of the interventionist will be given to the participants and they will be asked to contact the interventionist if they have any questions during the technique.

Physician will be available during the study period in the hemodialysis unite. In case of emergency cases during intervention period, the physician will perform assessment to the participants. Participants will be offered the appropriate treatment and medications according to the physician order and hospital strategy.

The control group:

A qualified nutritionist will run out a nutrition package session for hemodialysis patients in the control group. This nutrition package session will be for one session for one hour. This session will be conducted before dialysis session in a warm quite room with efficient light, temperature, and ventilation in the hemodialysis department.

Furthermore, the control group will be receiving the routine care at the hemodialysis unite during the study period. The patients will be receiving the routine care as follows: checking their vital signs, monitoring dialysis, reaction to the dialysis treatment and medication from the beginning to the end of the dialysis, and reviewing their medication and lab data. Furthermore, their medications and conditions will be evaluated and changed based on the physician's recommendation.

To prevent bias, the control group will not be offered any information about Benson relaxation technique during the study period. However, they are put on a waiting-list to receive the intervention after the active treatment group does. After the study period, the interventionist will perform the Benson relaxation technique to the control group. The training sessions will be conducted before dialysis session in a warm quite room with efficient light, temperature, and ventilation in the hemodialysis department. The interventionist will explain the technique verbally and a video of Benson relaxation technique will be displayed to participants. The technique will be repeated if necessary over one or two training sessions until the interventionist confirm that the participants in the control group acquired sufficient skills. Also, a Compact disc (CD) of Benson relaxation technique and handouts copies on how to elect Benson relaxation technique will be offered to the control group.

Physician will be available during the study period in the hemodialysis unite. In case of emergency cases during intervention period, the physician will perform assessment to the participants. Participants will be offered the appropriate treatment and medications according to the physician order and hospital strategy.

Planning for Data Analysis:

Descriptive and inferential statistics will be used to answer the research questions of this study. Exploratory data analysis (EDA) will be carried out to determine the normality of data. The raw data will be checked for normality distribution by using the Skewness and Kurtosis as well as Smirnov-Kolmogrov tests. Equality of variances will be checked for all variables using Levine's test.

Descriptive statistics will be conducted with presenting frequencies, percentages, median, range, means and standard deviations for the socio demographic variables among hemodialysis patients in Amman governmental Jordanian hospitals. Frequencies and percentages will be used to present the categorical variables. Moreover, Continuous variables will be described using the central tendency measures (means, and medians), the dispersion measures (standard deviation), and inter-percentile measures (P25, P50, and P75).

Inferential statistics as well as measures of central and dispersion the paired t test, analysis of variance for repeated measures, post hoc tests of S-N-K, Duncan, Scheffe and Tukey will be used to analyze data.

Characteristics of the study's participants will be compared between groups using the chi-square test for categorical variables and the t-test for continuous variables analysis to compare groups on demographic variables. After assessing the basic assumptions of the parametric tests; linearity, independence, homoscedasticity, and normality an Independent-t test will be used to compare the study's variables at baseline between two groups. Furthermore, Paired-sample t-test and repeated-measure analysis of variance (ANOVA) will be used to assess the effectiveness of the Benson relaxation technique intervention on the main outcome measure over time for both within and between study groups.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients who agree to participate in the study (by consent form).
* Hemodialysis patients begin alert, conscious, and oriented.
* Hemodialysis patients able to read and write in Arabic.
* Haemodialysis patients aged 18 years and above, participants of this age and above are adults and able to understand the items in the questionnaires in order to be able to answer them.
* Haemodialysis patients being on haemodialysis for at least six months and currently receiving haemodialysis at a minimum of two times per week. By 6 months, the routine for the hemodialysis procedure is established, and two times per week is the minimum number for dialysis sessions.

Exclusion Criteria:

* Hemodialysis patients with physical disability and physical limitation for learning and performing the Benson relaxation technique.
* Peritoneal dialysis or a kidney transplant patients.
* Patients who are taking antidepressants medication.
* Haemodialysis patients with cognitive impairment or mental health issues.
* Hemodialysis patients that face crisis intervention including changes in disease progress or loss of consciousness.
* Hemodialysis patients with emotional upheaval, such as death of a relative or a family member and divorce in their family, and those with any problems which had a negative impact on their mood during the previous month were excluded, The reason for these exclusions was that these complications might affect the concentration which is important in the relaxation technique and these patients might have difficulty in performing this procedure.
* No co-morbidity with other chronic disease like cancer, heart disease, etc. Diabetes and hypertension are included, because usually these co-morbidities are a part of renal failure; excluding them leads to limitation in generalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-02-14 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
The change of Pain level at baseline test (before intervention), a post-test (immediately after the intervention), and follow up at one month post-intervention, and follow up at two months' post-intervention. | at baseline test (before intervention), a post-test (immediately after the intervention), and follow up at one month post-intervention, and follow up at two months' post-intervention.
  Pain is the feeling of unpleasant sensory and discomfort which is experienced by hemodialysis patients. Pain will be measured by scores on the short form McGill Pain Questionnaire (SF-MPQ). The short form McGill Pain Questionnaire (SF-MPQ) consists of three parts:
  * The first part: consists of 15 descriptive adjectives, 11 sensory and four affective, which are rated on a four point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe), yielding three scores.
  * The second part: Visual Analogue Scale (VAS), which is a 10-centimeter horizontal line from 0 to 10 ranging from "no pain" to the "worst possible pain".
  * The third part: Present Pain Intensity (PPI), which is a six-point verbal rating scale on rating scale from 0 to 5, the words are: no pain (0), mild pain (1), discomforting (2), distressing (3), horrible (4), and excruciating (5).
The change of Perceived Stress Level at baseline test (before intervention), a post-test (immediately after the intervention), and follow up at one month post-intervention, and follow up at two months' post-intervention. | at baseline test (before intervention), a post-test (immediately after the intervention), and follow up at one month post-intervention, and follow up at two months' post-intervention.
  Perceived stress refers to an undesired state of feeling frustrated, anger and nervous of anxious, which is experienced by hemodialysis patients.
  The level of stress for the hemodialysis patients will be assessed using the Perceived Stress Scale. The perceived stress scale (PSS-10) has 10 items on a 5-point Likert scale (0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often). Four positively stated items (item 4, 5, 7, and 8) are reversely scored (0 = very often, 1 = fairy often, 2 = sometimes, 3 = almost never, 4 = never). The sum of the 10 items represents the total score, with higher scores representing higher levels of perceived stress. Individual scores on the Perceived stress score (PSS-10) can range from 0 to 40 with higher scores indicating higher perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Lam Soh, PhD, Study Director — Associate Professor at Department of Nursing and Rehabilitation at UPM

IPD SHARING:
Plan to Share IPD: Yes
all Information Participant data (IPD) that underlie results in a publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available within 6-8 months of study completion.
Access Criteria: Access criteria has not been decided yet.

REFERENCES:
- [Result] Mahdavi A, Gorji MA, Gorji AM, Yazdani J, Ardebil MD. Implementing Benson's Relaxation Training in Hemodialysis Patients: Changes in Perceived Stress, Anxiety, and Depression. N Am J Med Sci. 2013 Sep;5(9):536-40. doi: 10.4103/1947-2714.118917. PMID 24251271
- [Result] Heidari Gorji MA, Davanloo AA, Heidarigorji AM. The efficacy of relaxation training on stress, anxiety, and pain perception in hemodialysis patients. Indian J Nephrol. 2014 Nov;24(6):356-61. doi: 10.4103/0971-4065.132998. PMID 25484528
- [Result] Rambod M, Sharif F, Pourali-Mohammadi N, Pasyar N, Rafii F. Evaluation of the effect of Benson's relaxation technique on pain and quality of life of haemodialysis patients: a randomized controlled trial. Int J Nurs Stud. 2014 Jul;51(7):964-73. doi: 10.1016/j.ijnurstu.2013.11.004. Epub 2013 Nov 25. PMID 24332569
- [Derived] Abu Maloh HIA, Soh KL, Chong SC, Ismail SIF, Soh KG, Abu Maloh DI, Al Yateem N, AbuRuz ME. The Effectiveness of Benson's Relaxation Technique on Pain and Perceived Stress Among Patients Undergoing Hemodialysis: A Double-Blind, Cluster-Randomized, Active Control Clinical Trial. Clin Nurs Res. 2023 Feb;32(2):288-297. doi: 10.1177/10547738221112759. Epub 2022 Aug 1. PMID 35915917
- See also: Study aimed to evaluate the effect of Benson's Relaxation on depression, anxiety and stress in patients undergoing hemodialysis. — http://www.ijmrhs.com/abstract/the-effect-of-bensons-relaxation-on-depression-anxiety-and-stress-in-patients-undergoing-hemodialysis-6593.html